CLINICAL TRIAL: NCT07309484
Title: The Role of Lifestyle in Maintaining Health: Biological, Psychological and Social Responses of the Organism to Lifestyle
Brief Title: Lifestyle and Its Association With Maintaining Health
Acronym: LifeHealth-OBS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Zadar (Other)
Collaborators: General Hospital Zadar (Other); Agricultural, Food and Veterinary School Stanko Ožanić, Zadar, Croatia (Unknown); University of Primorska (Other); University of Cadiz (Other); University of Camerino (Unknown); International Hellenic University (Other); University of Split, School of Medicine (Other); Andrija Stampar Teaching Institute of Public Health (Unknown)
Responsible Party: Principal Investigator, Marija Ljubičić, Assistant Professor, PhD, Department of Health Studies, University of Zadar, Croatia, University of Zadar
Other Study IDs: IP UNIZD 2025-27040_obs; EU Next Generation NPOO (Other Grant/Funding Number: European Union / Sveučilište u Zadru)
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Lifestyle (Sedentary Behavior and Physical Activity); Mental Health; Nutrition; Sleep; Stress; Unhealthy Diet, Exercise, Smoking, and Alcohol Use; Body Mass Index
Keywords: Lifestyle; stress; nutrition; sleep; depression; anxiety; smoking; physical activity; Mediterranean Diet; social relationship; attitude
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being; Smoking; Alcohol Drinking; Depression; Anxiety Disorders; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group includes approximately 2500 respondents from European Union: This group includes approximately 500 respondents from each of five Mediterranean European Union countries: Croatia, Greece, Italy, Slovenia, and Spain. Participants are adults who will complete an online questionnaire on lifestyle habits, diet, physical activity, sleep, stress perception, mental health, social relationships, and overall health. The aim is to describe current lifestyle patterns and examine how these habits relate to physical and mental health in Mediterranean populations. Participation is voluntary, and respondents can withdraw at any time.

SUMMARY:
This study is part of the LIFEHEALTH project and will be carried out in five Mediterranean European Union countries: Croatia, Greece, Italy, Slovenia, and Spain. The aim of this study is to assess adults' lifestyle habits and how they relate to their physical and mental health. Respondents in each country will be invited to complete an online questionnaire. The survey will ask about consumption of the Mediterranean diet, physical activity, sleep habits, stress perception, mental health, social relationships, and overall health. Each country will include about 500 participants to ensure a representative sample of adults living in Mediterranean regions.The questionnaire will be translated into local languages and participation is voluntary. Multiple linear or logistic regresion wil be used to assess relation between variables. These analyses will help identify which factors are most strongly linked to health outcomes. The results of this study will help researchers describe current lifestyle patterns in the Mediterranean population. They will also examine how different lifestyle habits are linked to physical and mental health. The findings may support public health initiatives and help plan future research to improve health and well-being.

DETAILED DESCRIPTION:
This study is part of the LIFEHEALTH project and will be conducted in five Mediterranean European Union countries: Croatia, Greece, Italy, Slovenia, and Spain. The study is planned for the first year of the project and aims to assess adults' lifestyle habits and their relationship to physical and mental health.

Each participating country will recruit approximately 500 respondents, selected to provide a representative sample of adults living in Mediterranean regions. Inclusion criteria are: adults aged 18 years or older, residing in the participating country, and willing to complete an online questionnaire. There are no specific exclusion criteria, except inability to provide informed consent or complete the survey.

Data will be collected via an online questionnaire. The survey includes questions about: consumption of the Mediterranean diet, physical activity, sleep habits, stress perception, mental health, social relationships, overall health. The questionnaire will be prepared in English and translated into local languages using the back-translation method to ensure accuracy and consistency. Each country's team will distribute the survey using digital platforms such as email, WhatsApp, and other online tools. Participation is voluntary, and respondents will be informed about the study objectives, procedures, and their rights before completing the questionnaire. Respondents may withdraw at any time without consequence. Before starting the survey, respondents will click the "I Agree" button to show that they understand the study and agree to take part. Statistical analyses will examine relationships between lifestyle factors and self-reported physical and mental health. The analyses will help identify lifestyle habits most strongly associated with health outcomes across countries. The collected data and results interpretation will provide a detailed overview of current lifestyle patterns in Mediterranean populations and its asociations between lifestyle and health outcomes. The findings will inform public health initiatives and support planning of future research aimed at improving health and well-being .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Residents of participating European countries
* Access to the internet
* Ability to provide informed consent
* Completion of the online questionnaire

Exclusion Criteria:

* Individuals under 18 years of age
* Non-residents of the participating European countries
* Inability to understand the language of the questionnaire
* Cognitive and/or technical difficulties preventing completion of the online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this cross-sectional study, participants from selected European Union countries will complete an online questionnaire covering key aspects of health, dietary habits, physical activity, mental health, and socioeconomic factors. Participants will be recruited from healthcare and educational institutions, fitness centers, online platforms, workplaces, associations, as well as through advertising materials and media outreach.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mediterranean diet adherence | through study completion, an average of 1 year
  Assessed using validated dietary questionnaires to evaluate participants' adherence to Mediterranean diet principles and monitor changes over time.
  The Mediterranean Dietary Serving Score (MDSS) evaluates 14 food groups, including cereals, fruits, vegetables, olive oil, nuts, dairy, meat, fish, eggs, legumes, potatoes, wine/beer, and sweets. Consumption is rated on a 7-point Likert scale. Scores above 14 indicate regular adherence to a Mediterranean diet.
Physical Activity | through study completion, an average of 1 year
  Assessed using the Godin Leisure-Time Exercise Questionnaire to evaluate participants' frequency and intensity of physical activity during free time, and to monitor changes in exercise behavior over time.
  Godin Leisure-Time Exercise Questionnaire (GLTEQ), calculates a total score by multiplying the weekly frequency of strenuous, moderate, and light activities by 9, 5, and 3, respectively. Higher scores indicate greater levels of physical activity and allow monitoring of changes in exercise behavior over time.
Sleep Hygiene | through study completion, an average of 1 year
  Assessed using validated sleep hygiene questionnaires to evaluate participants' sleep habits, routines, and behaviors that promote restorative sleep.
  The Sleep Hygiene Index (SHI) consists of 13 items for self-assessment of sleep-related behaviors. Participants rate how often they engage in specific behaviors on a 5-point scale: 0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always. Scores are summed to provide a global sleep hygiene score, with higher scores indicating poorer (maladaptive) sleep hygiene and a greater presence of behaviors that disrupt sleep quality
Perceived Stress | through study completion, an average of 1 year
  Self-reported questionnaire to assess perceived stress levels. The Perceived Stress Scale-10 (PSS-10) assesses the perception of stressful situations over the past month through 10 items rated on a 0-4 scale. Total scores range from
Attitudes toward a Healthy Lifestyle | through study completion, an average of 1 year
  The Attitudes toward a Healthy Lifestyle Questionnaire is based on six core domains of lifestyle medicine: balanced nutrition, regular physical activity, effective stress management, sleep quality, quality of interpersonal relationships, and avoidance of risky behaviors such as smoking and alcohol consumption. The instrument consists of 15 items. Responses are recorded using a 5-point Likert scale, where 1 indicates complete disagreement and 5 indicates complete agreement with the statement. Reverse scoring is applied to negatively worded items (items 1, 4, 7, 8, 10, and 12). The total scale score is calculated by summing the responses to all items, resulting in a possible score range from 15 to 75. Higher total scores reflect more positive attitudes toward a healthy lifestyle.
Healthy Days (Physical and Mental Health) | through study completion, an average of 1 year
  Assessed using the CDC Healthy Days questionnaire to evaluate the number of days in the past 30 days when participants perceived their physical or mental health as not good.
  The Health Related Quality of Life 14 item measure (CDC HRQOL 14) is a generic self report questionnaire developed by the U.S. Centers for Disease Control and Prevention to assess overall health related quality of life. It comprises 14 items that capture perceived physical and mental health status over the past 30 days, including self rated general health, the number of days with poor physical health, poor mental health, days when health limited usual activities, and additional questions on activity limitations and symptoms such as pain, depression, anxiety, rest, and energy. The measure provides a summary of health related quality of life and has been widely used in public health surveillance, research, and population health studies. Higher scores generally reflect poorer health related quality of life.
Personal Wellbeing | through study completion, an average of 1 year
  Personal Wellbeing Index (PWI) is self-report measuring subjective well-being across seven domains: standard of living, health, achieving in life, personal relationships, personal safety, community-connectedness, and future security. Each domain is rated on an 11-point Likert scale (0-10), with higher scores indicating greater subjective well-being. The total PWI score is calculated as the mean of the domain scores.

SECONDARY OUTCOMES:
Association between lifestyle habits and physical health | through study completion, an average of 1 year
  Relationship between lifestyle factors and self-reported physical health status
Association between lifestyle habits and mental health | through study completion, an average of 1 year
  Relationship between lifestyle factors and self-reported mental health and stress perception.
Sociodemographic and health-related characteristics | through study completion, an average of 1 year
  Sociodemographic, health, and anthropometric characteristics of respondents across participating countries.
Associations between lifestyle domains and body mass index. | through study completion, an average of 1 year
  To assess attitudes toward a healthy lifestyle and to explore their relationships with specific lifestyle domains, including nutrition, physical activity, sleep, stress management, interpersonal relationships, sociodemographic characteristics, and body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Marija Ljubičić, Principal Investigator — University of Zadar, Croatia
Locations (1):
- University of Zadar, Zadar, Croatia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and compliance with GDPR regulations protecting participants' personal information."